CLINICAL TRIAL: NCT03321747
Title: Phase I/II Trial Evaluating Five Fraction SABR Dose Escalation for Early Stage Squamous Cell Carcinoma of the Lung
Brief Title: Five Fraction SABR Dose Escalation for Early Stage Squamous Cell Carcinoma of the Lung
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: After completion of Phase I, it was decided not to initiate Phase II of the study.
Sponsor: Indiana University (Other)
Collaborators: Indiana University School of Medicine (Other)
Responsible Party: Principal Investigator, Tim Lautenschlaeger, Assistant Professor of Radiation Oncology, Indiana University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IUSCC-0624
Record Dates: First submitted 2017-10-23; First posted 2017-10-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: This trial is a Phase I/II study designed to determine the maximum tolerated radiation dose and evaluate the efficacy of dose escalated SABR for early stage lung squamous cell carcinoma.
  *The Phase l portion of this study was completed. However; the trial will not continue into Phase II as originally planned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (5):
- Phase 1/Dose Level 1 (Experimental): 11 Gy will be given in 5 fractions for a total dose of 55 Gy
  Interventions: Radiation: Stereotactic Ablative Body Radiation (SABR)
- Phase 1/Dose Level 2 (Experimental): 12 Gy will be given in 5 fractions for a total dose of 60 Gy
  Interventions: Radiation: Stereotactic Ablative Body Radiation (SABR)
- Phase 1/Dose Level 3 (Experimental): 13 Gy will be given in 5 fractions for a total dose of 65 Gy
  Interventions: Radiation: Stereotactic Ablative Body Radiation (SABR)
- Phase 1/Dose Level 4 (Experimental): 14 Gy will be given in 5 fractions for a total dose of 70 Gy
  Interventions: Radiation: Stereotactic Ablative Body Radiation (SABR)
- Phase 2 (Experimental): The maximum tolerated radiation dose determined during Phase 1 (i.e. 11, 12, 13, or 14 Gy) will be given in 5 fractions for a total dose of 55, 60, 65, or 70 Gy.
  Interventions: Radiation: Stereotactic Ablative Body Radiation (SABR)

INTERVENTIONS:
Radiation: Stereotactic Ablative Body Radiation (SABR) — Treatments shall not be delivered more frequently than every other day.

SUMMARY:
The purpose of this study is to test whether 5 fraction stereotactic ablative body radiation (SABR) is safe and improves local control for early state squamous cell carcinoma of the lung. While three fraction SABR is effective for the treatment of early stage non small cell lung carcinoma (NSCLC) of all histologies, it is not safe for many patients. While four and five fraction SABR is safe, recently published data and our institutional data suggests that local control for early stage squamous cell carcinoma of the lung using the current four or five fraction SABR is suboptimal.

DETAILED DESCRIPTION:
1. Primary Objectives During Phase I study - Determine the safety and maximum tolerated radiation dose for five fraction SABR for squamous cell cancer of the lung.

   During Phase II study - Determine 2 year local control of dose escalated five fraction SABR vs. institutional historical control standard dose SABR in squamous cell cancer of the lung.
2. Phase II Secondary Objectives

   * Determine overall survival, progression free survival and patterns of failure after SABR.
   * Determine tolerability of dose escalated SABR.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥ 18 at time of consent.
2. Ability to provide written informed consent and HIPAA authorization.
3. Pathological diagnosis of squamous cell carcinoma of the lung.
4. Staging PET/CT (invasive mediastinal staging strongly encouraged but not required).
5. Tumors < 7cm
6. Any location eligible for SBRT (including, but not limited to, peripheral, chest wall abutting and central tumors)
7. N0 M0 disease
8. Plan to undergo four or five fraction SABR
9. Baseline PFTs available within 6 months of treatment start or will be obtained prior to treatment start (no finding will exclude patient from enrollment in trial)

Exclusion Criteria

1. Previous radiation therapy to the lung per investigator discretion.
2. Inability to comply with treatment per investigator discretion.
3. Inability to follow standard of care follow up recommendations per investigator discretion.
4. KPS<40

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2020-07-09 (Actual); Study Completion 2020-07-09 (Actual)

PRIMARY OUTCOMES:
Rate of dose limiting toxicities (DLTs) in each cohort during Phase 1 | 30 days
  Any event per CTCAE v.4 that occurs within 30 days from the start of SABR, and is possibly, probably or definitely related to treatment, and is related to a specific list of symptoms which are outlined in the protocol.

SECONDARY OUTCOMES:
Local control during Phase 2 | 2 years
  Failures will be classified as local failures if failing within or immediately adjacent to the PTV, unless judged by the investigator team to convincingly be a separate lesion from the treated lesion (i.e. new lesion within a planning target volume but across a fissure).
Overall survival | 2 years
  Length of time start of treatment that patients are still alive

CONTACTS AND LOCATIONS:
Overall Officials: Tim Lautenschlaeger, MD, Principal Investigator — Indiana University
Locations (3):
- United States (3):
  - Indiana University Health Hospital, Indianapolis, Indiana
  - Indiana University Health Methodist Hospital, Indianapolis, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No